CLINICAL TRIAL: NCT00970021
Title: Use of the Medicinal Mushroom Agaricus Blazei Murill in Addition to High Dose Chemotherapy in Patients With Multiple Myeloma.
Brief Title: Agaricus Blazei Murill in Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Responsible Party: Principal Investigator, Jon Magnus Tangen, Senior Consultant, Oslo University Hospital
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Ando-01
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2014-02-25 (Estimated); Status verified 2014-02

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Water

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Water with artificial colour (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Intake of 60 ml placebo daily in addition to chemotherapy
- Extract of agaricus blazei Murill (Active Comparator): Agaricus blazei Murill
  Interventions: Dietary Supplement: Intake of 60 ml agaricus daily in addition to chemotherapy

INTERVENTIONS:
Dietary Supplement: Intake of 60 ml placebo daily in addition to chemotherapy — The patients will drink 60 ml of placebo daily from start of stem cell mobilizing treatment until one week after the end of aplasia after high dose melphalan. Duration of treatment is approximately 7 weeks.
  Other Names: Water with artificial colour
  Arms: Water with artificial colour
Dietary Supplement: Intake of 60 ml agaricus daily in addition to chemotherapy — The patients will drink 60 ml of agaricus extract from the start of stem cell mobilizing treatment until one week after the end of aplasia after high dose melphalan. Duration of treatment: Approximately 7 weeks
  Other Names: Commercial name: AndoSan(TM)
  Arms: Extract of agaricus blazei Murill

SUMMARY:
Extract from the mushroom Agaricus blazei Murill har been shown to have strong immunomodulating properties both in cell cultures, animal models and in humans. Furthermore antitumor properties have been shown in animal models, among them in mice with multiple myeloma. The investigators now want to investigate the effect of Agaricus as supplementary treatment in addition to chemotherapy in patients with multiple myeloma.

DETAILED DESCRIPTION:
Patients who are scheduled to undergo high dose chemotherapy for multiple myeloma will receive in addition in a double blinded manner 60 ml of agaricus extract or placebo once daily from the start of stem cell mobilizing therapy until one week after the end of aplasia after high dose melphalan.

Primary endpoints will be cytokine levels of degree of activation of tumor supressor genes before and after start of the investigational product.

Secondary endpoints will be treatment response and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled to undergo high dose chemotherapy with autologous stem cell support for multiple myeloma

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Cytokine levels in serum | 7 weeks

SECONDARY OUTCOMES:
Quality of Life | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jon-Magnus Tangen, Principal Investigator — Department of Hematology, Oslo University Hospital, Ulleval
Locations (1):
- Department of hematology, Oslo University Hospital, Ullevaal, Oslo, Norway

REFERENCES:
- [Derived] Tangen JM, Tierens A, Caers J, Binsfeld M, Olstad OK, Troseid AM, Wang J, Tjonnfjord GE, Hetland G. Immunomodulatory effects of the Agaricus blazei Murrill-based mushroom extract AndoSan in patients with multiple myeloma undergoing high dose chemotherapy and autologous stem cell transplantation: a randomized, double blinded clinical study. Biomed Res Int. 2015;2015:718539. doi: 10.1155/2015/718539. Epub 2015 Jan 18. PMID 25664323